CLINICAL TRIAL: NCT00729274
Title: HYPERTONIC SALINE IN ACUTE VIRAL BRONCHIOLITIS: A RANDOMIZED CLINICAL TRIAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was not approved by funding organization
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre de Recheche du Centre Hospitalier Université Laval (Other)
Responsible Party: Dr. Chantal Guimont MD, PhD, Pediatric Research Unit of Laval University Hospital Center.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 222207
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Acute Viral Bronchiolitis.
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypertonic saline solution (Active Comparator): Hypertonic Saline 3% solution alone.
  Interventions: Drug: normal saline solution
- nebulized normal saline solution (Placebo Comparator): 2 nebulisation with 30 minute interval (max 4ml)
  Interventions: Drug: normal saline solution

INTERVENTIONS:
Drug: normal saline solution — Two 4ml nebulizations with 30 minute interval
  Other Names: Physiologic saline solution

SUMMARY:
The purpose of this study is to determine whether nebulized hypertonic saline solution reduces the admission rate 48 hours after initial treatment in the emergency department, when compared to normal saline solution (placebo). We hypothesise that patients with bronchiolitis who receive nebulized hypertonic saline solution will have less respiratory distress, less duration of symptoms and therefore less risk of being hospitalized than those receiving normal saline solution.

DETAILED DESCRIPTION:
Acute viral bronchiolitis is the principal lower respiratory tract infection in infants worldwide, 10% of canadian infants are affected each year. It is characterized by a first episode of difficulty to breathe, preceded by symptoms of fever, rhinorrhea and cough. The only accepted treatment for bronchiolitis is nasal cleaning, hydration and oxygen administration. Multiple studies have documented variation in diagnostic testing, clinical scores used and different treatment modalities. This suggests a lack of consensus on the diagnosis, on criteria for hospitalization and on treatment. Nebulized 3% hypertonic saline solution has been proposed as a potential treatment for the reduction in the severity of respiratory symptoms and the rate of admission in bronchiolitis, it has never been studied alone and the effect on the rate of admission has been little studied.

We propose a randomized double blind multicenter clinical trial on infants 6 weeks to 12 months old with moderate or severe bronchiolitis, in 9 emergency departments of hospitals situated in different provinces across Canada, during 3 winter seasons. We hypothesise that infants with bronchiolitis treated with nebulized hypertonic 3% saline solution would have less risk of being hospitalized and would have shorter and less intense respiratory symptoms than those infants treated with nebulized normal saline solution. Our principal objective is to determine if nebulized 3% hypertonic saline solution reduces admission rate 48 hours after treatment compared to placebo. Secondary objectives are to compare between groups intensity of respiratory symptoms measured by different clinical scores (RDAI,PRAM, PASS and IRAS), duration of symptoms, length of hospital stay, added secondary effects and subsequent office visits for the same problem.

Comparatively to other therapies already studied such as (dexamethasone and epinephrine), hypertonic 3% saline constitutes an interesting choice due to the absence of potential secondary effects. Our study will try to optimize the utilization of hospital resources involved in the treatment of bronchiolitis. Infants suffering from this disease could therefore profit from better treatments which will be reflected in a better condition, life quality and consequently those of their parents.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of viral bronchiolitis
* Age 6 weeks to 12 months
* Clinical Score IRAS >3 and <8

Exclusion Criteria:

* prematurity <30 weeks
* younger than 6 weeks of age
* chronic lung disease
* immunosuppression.
* History of wheezing or asthma.
* Clinical Score IRAS >9
* parents refuse study

Ages: 6 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Hospitalization Rate | After 48 hours of treatment in the emergency department

SECONDARY OUTCOMES:
The IRAS (Infant Respiratory Assessment Score) will be measured after each Treatment to verify improvement. | 30 minutes after each nebulization

CONTACTS AND LOCATIONS:
Overall Officials: Guimont Chantal, MD, PhD., Principal Investigator — Laval University Hospital Center, Quebec, Canada.
Locations (1):
- Laval University Hospital Center, Québec, Quebec, Canada